CLINICAL TRIAL: NCT01674101
Title: A Pilot Study on the Effects of Preoperative Physical Therapy in Adolescents and Young Adults Diagnosed With a Lower Extremity Malignancy
Brief Title: Effects of Preoperative Physical Therapy in Patients With Lower Extremity Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Tennessee Physical Therapy Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PTSARC; TPTA (YR 1) (Other: Tennessee Physical Therapy Association); NCI-2012-01920 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Osteosarcoma; Ewing's Sarcoma; Rhabdomyosarcoma; Synovial Sarcoma; Malignant Peripheral Nerve Sheath Sarcoma; Malignant Fibrous Histiocytoma of the Bone; Chondrosarcoma of the Bone
Keywords: Lower extremity malignancy
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma, Synovial | interventions — Physical Therapy Modalities; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical Therapy (Experimental): The intervention group will receive PT 3 times per week for 60 minutes each session. The therapy sessions will include endurance, strengthening, and stretching exercises.
  Exercise time and resistance will be progressed per individual's medical status and per participant's tolerance. All participants will be given a tailored home exercise program (HEP).
  Participants will participate in PT 10 weeks prior to surgery and 10-12 weeks after surgery. Subjects will be seen by the physical therapist both when inpatient and outpatient. Patients will not be seen for PT if platelet count is less than 20,000mm3 and/or hemoglobin is less than 8g/dL.
  Interventions: Other: Endurance; Other: Strengthening; Other: Stretching; Other: Home exercise program

INTERVENTIONS:
Other: Endurance — Endurance exercise will consist of ambulating with assistive devices as needed, upper extremity (UE) ergometer, and/or playing the Wii.
  Other Names: Physical therapy
Other: Strengthening — Strengthening exercises will involve both UE's and LE's. For UE's, bicep curls, triceps curls, shoulder flexion, and/or press-ups from the therapy mat or wheelchair will be included. For the LE's, bridging, long arc quads, hamstring curls, calf raises in standing, single LE squats, and/or dorsiflexion (DF) in supine will be performed on the uninvolved extremity.
  Other Names: Physical therapy
Other: Stretching — Stretching will consist of ankle stretch into DF in supine or long sitting, hamstring stretch in supine with hip flexed to 90 degrees, and trunk extension in sitting.
  Other Names: Physical therapy
Other: Home exercise program — All participants will be given a tailored home exercise program (HEP) including endurance exercises, strengthening, and stretching exercises to be completed on days they do not have PT. If the participants return home, they will be asked to complete the HEP at least 3 days per week. The physical therapist will contact the participant weekly to modify the HEP if necessary and determine compliance.
  Other Names: Physical therapy

SUMMARY:
This application proposes a prospective clinical trial to evaluate the impact of adding a focused physical therapy (PT) intervention to the preoperative regimen of individuals diagnosed with a malignancy of the lower extremity (LE). The primary aim will be to determine if individuals diagnosed with a malignancy of the LE can participate in a 10 week preoperative strengthening, stretching, and aerobic exercise regimen.

DETAILED DESCRIPTION:
The intervention group will receive PT 3 times per week for 60 minutes each session. The therapy sessions will include endurance, strengthening, and stretching exercises. Endurance exercises will consist of ambulating with assistive devices as needed, using the upper extremity (UE) ergometer, and/or playing the Wii. Strengthening exercises will involve both UE's and LE's. For UE's, bicep curls, triceps curls, shoulder flexion, and/or press-ups from the therapy mat or wheelchair will be included. For the LE's, bridging, long arc quads, hamstring curls, calf raises in standing, single LE squats, and/or dorsiflexion (DF) in supine will be performed on the uninvolved extremity. Resistance and exercise time will be increased depending upon participant's tolerance. Stretching will consist of ankle stretch into DF in supine or long sitting, hamstring stretch in supine with hip flexed to 90 degrees, and trunk extension in sitting.

PRIMARY OBJECTIVE

To determine if individuals diagnosed with a malignancy of the LE can participate in a 10 week preoperative strengthening, stretching, and aerobic exercise regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient being treated at St. Jude Children's Research Hospital
* Permission from participant's physician
* Participants must be between the ages of 6 and 30 years of age
* Patient is newly diagnosed with LE malignancy as shown by biopsy. Diagnoses include: osteosarcoma, Ewing's sarcoma, rhabdomyosarcoma, synovial sarcoma, malignant peripheral nerve sheath sarcoma, malignant fibrous histiocytoma of the bone and chondrosarcoma of the bone, or any other LE malignancy that requires surgical intervention.
* Patient has Karnofsky score ≥ 50 or WHO/ECOG ≤ 2 if ≥ 16 years of age
* Lansky score ≥ 50 for patients age < 16
* Surgical intervention is planned primary mechanism of local control
* Negative pregnancy test
* All patients and/or their parents or legal guardians must sign a written informed consent

Exclusion Criteria:

* Patients with serious, non-healing wound, ulcer or bone fracture (other than pathologic fracture)
* Pre-morbid condition that prevents patient from ambulating
* Patients who do not have at least 10 weeks before receiving local control

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of a 10 week physical therapy intervention program | Up to 12 weeks post surgery
  Determine if individuals diagnosed with a malignancy of the LE can participate in a 10 week preoperative strengthening, stretching, and aerobic exercise regimen. We will consider the study to be feasible if at least 60% of the patients are able to complete at least 50% of their scheduled PT sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M. Corr, PT, DPT, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols